CLINICAL TRIAL: NCT06317506
Title: Assessment of Methylation Pattern Related to Pain Sensation in Children With Intellectual Disability: a Cross-sectional Study
Brief Title: Methylation Pattern and Pain Sensation in Children With Intellectual Disability
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 43/2022
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Intellectual Disability
Keywords: Pain; Intellectual disability; Epigenetics
MeSH Terms: conditions — Intellectual Disability; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with ID: The presence of intellectual disability will be evaluated according to DSM-V criteria
- Children without ID: The presence of intellectual disability will be evaluated according to DSM-V criteria

SUMMARY:
Previous literature data indicate that children with intellectual disability (ID) experience more severe pain and more frequently than their cognitively healthy peers, during their daily life. Repeated and chronic pain exposure triggers a vicious circle of hyperalgesia and reduction of the impaired cognitive and adaptive function. Furthermore, these children are unable to rationalize any intervention targeted to contain potentially painful actions.

Epigenetics studies mechanisms responsible for a set of modifications that regulate gene expression without altering the DNA sequence itself. DNA methylation and posttranslational modification of histones are the main epigenetic mechanisms. It is widely accepted that these mechanisms can be engaged by environmental experience, such as early life trauma, pain or addiction leading to the idea of epigenetics as 'a bridge' between genes and environment.

Several epigenetic studies evaluated genes coding proteins involved in recycling of neurotransmitters (SCL6A4), in transmission of painful stimuli (TRPA1) and in response to analgesics (OPRM1). In particular, some studies assessed TRPA1 gene, coding for a cationic channel responsible for the transmission of thermal-painful sensations, and SCL6A4, a serotonin-recycling transmembrane protein presents at inter-synaptic level, have highlighted the importance of methylation in a pathological experience of chronic pain and anxiety disorder in the adult population. Opioid receptor OPRM1 is involved in the endogenous and exogenous opioid-mediated analgesia and a recent work in a group of adolescents treated for idiopathic scoliosis highlights a link between greater pain post-surgery and methylation of this gene. In this context, children with ID are at greater risk of undertreatment both for the difficulty in pain recognition and for the fear of medication-adverse reactions.

The epigenetic study of the aforementioned genes in children with ID associated with an evaluation of painful experiences and clinical history, could help understanding a scenario that it is still complex nowadays before the eyes of parents and caregivers and healthcare workers.The finding of a different methylation pattern in children with ID could in part explain the different pain experience.

ELIGIBILITY:
Inclusion Criteria:

- Children with scheduled venipuncture or venous cannulation for diagnostic or therapeutic reasons, with and without severe intellectual disability.

Exclusion Criteria:

- Presence of Autism spectrum disorder (ASD) according to DSM-V criteria.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with intellectual disabilities and healthy controls recruited:
  * at the Pediatric Department, general and surgical Day-hospital, Child Neuropsychiatry service and Pediatric Emergency Department of the IRCSS Burlo-Garofolo, Trieste, Italy;
  * at the Pediatric Department of "Santa Maria degli Angeli" Hospital, in Pordenone, Italy;
  * at the Pediatric Department of Monfalcone Hospital, in Monfalcone, Gorizia, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Between groups differences in methylation levels | Through study completion, an average of 18 months
  Evaluation of differences in methylation levels of three genes promoters (SCL6A4, OPRM1, TRPA1) in children with severe intellectual disability in comparison with their cognitively healthy peers

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy